CLINICAL TRIAL: NCT04044274
Title: Evaluation of a Novel Method for Increasing Intraocular Pressure in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv.-Doz. Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-120219
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IOPstim (Experimental)
  Interventions: Device: IOPstim; Device: Suction Cup

INTERVENTIONS:
Device: IOPstim — IOPstim (IMEDOS, Jena, Germany) is a device exerting defined pressure to the sclera and hence increasing IOP.
Device: Suction Cup — Suction Cup is a device exerting defined suction to the clear and hence increasing IOP

SUMMARY:
Adequate perfusion is necessary for maintaining tissue function. This applies also for the eye, in which ocular perfusion pressure (OPP) is generally estimated as the difference between mean arterial pressure (MAP) and intraocular pressure (IOP). In the latter formula, IOP substitutes for central retinal venous pressure (CRVP), which is assumed to be slightly higher than IOP to allow blood flow to exit the eye. It has, however, been found that in some patients CRVP is elevated and significantly higher than IOP, which would lead to a decrease in OPP which is not taken in account with the proposed formula. Therefore, techniques for measurement of CRVP are warranted. Recently, a new, method for measurement of this parameter without corneal contact has been introduced. Briefly, with this method, IOP is elevated until the vein collapses, which then equals CRVP. In the present study this technique will be applied in 12 healthy subjects to validate whether the values that are preset by the device correlate to measurements obtained with standard Goldmann applanation tonometry. For this purpose, IOP will be experimentally increased in steps of approximately 5mmHg until it reaches 40mmHg as measured by applanation tonometry. After a resting period of 30 minutes, IOP will be again increased stepwise to 40 mmHg while retinal vessel diameters will be monitored using dynamic vessel analyzer. During this session CRVP will be measured. After another resting period of 30 minutes IOP will be stepwise increased a third time and after each step OCT, OCT-A and OCT EDI will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years
* Non-smokers
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 1 Dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug (except contraceptives)
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks
* Pregnancy, planned pregnancy or lactating

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | 15 Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhöfer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria